CLINICAL TRIAL: NCT02320162
Title: "School-based Oral Health Education Program Using Experiential Learning or Traditional Lecturing in Children and Adolescents: a Clinical Trial"
Brief Title: School-based Oral Health Education Program Using Experiential Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matina Angelopoulou (Other)
Responsible Party: Sponsor-Investigator, Matina Angelopoulou, Assistant Professor, Marquette University
Organization: Marquette University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Marquette U
Record Dates: First submitted 2014-12-11; First posted 2014-12-19 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2014-12

CONDITIONS: Caries; Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Experiential learning (Experimental): Oral health education using experiential learning (EL)
  Interventions: Behavioral: Experiential learning oral health education
- Traditional lecturing (Placebo Comparator): Oral health education using traditional lecturing (TL)
  Interventions: Behavioral: Experiential learning oral health education

INTERVENTIONS:
Behavioral: Experiential learning oral health education

SUMMARY:
The aim of this project was to compare the effectiveness of experiential learning (EL) and traditional lecturing (TL) school-based oral health education on the oral health knowledge, attitude, habits, oral hygiene, gingival health and caries incidence of 10 and 13-year-old Greek children. Thee hundred and fifty children were selected from three areas of Greece. Information on oral health knowledge, attitude and behaviour were obtained using a questionnaire. Dental plaque was recorded using a modified hygiene index, gingivitis was assessed using the simplified gingival index and dental caries was measured by recording the number of Decayed, Missing and Filled teeth (DMFT) using the British Association for the Study of Community Dentistry (BASCD) criteria. All children were examined by two calibrated dentists, using a World Health Organisation (WHO) periodontal probe and artificial light. Questionnaires were delivered and clinical examinations were performed at baseline and at 6 and 18 months post-intervention. The EL oral health educational program was implemented by teachers using the program's manual.

ELIGIBILITY:
Inclusion Criteria:

* 10 and 13 year-old children
* For the EL group, students were recruited from schools that had teachers previously trained in EL
* Students recruited for the TL group attended schools of the same geographical location as students in the EL group

Exclusion Criteria:

* Contributory medical history

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 351 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in dental plaque, gingivitis and caries at 6 and 18 months in 350 children | baseline, 6 and 18 months
  350 children were clinically examined and dental plaque, gingivitis and caries were recorded using appropriate indexes. 6 and 18 months later, children were re-examined using the same method to test if there was any change on the dental plaque, gingivitis and caries level and if this change differ significantly between the two different oral health education groups (Experiential learning or Traditional Lecturing).

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Oulis, DDS,MS,PhD, Study Chair — Dental School, University of Athens

REFERENCES:
- [Derived] Angelopoulou MV, Kavvadia K, Taoufik K, Oulis CJ. Comparative clinical study testing the effectiveness of school based oral health education using experiential learning or traditional lecturing in 10 year-old children. BMC Oral Health. 2015 Apr 28;15:51. doi: 10.1186/s12903-015-0036-4. PMID 25924670